CLINICAL TRIAL: NCT02359942
Title: The Effect of Citric Acid as the Test Meal on the Diagnostic Accuracy of the 13C-Urea Breath Test in Korean, Randomized Controlled, Open Label Prospective Study
Brief Title: The Diagnostic Validity of the Urea Breath Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Purpose: Diagnostic
Other Study IDs: B-1412/279-004
Record Dates: First submitted 2015-01-18; First posted 2015-02-10 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; Eradication; Urea breath test
MeSH Terms: interventions — Citric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citric acid group (Experimental): Giving the citric acid (4g) as test meal before UBT
  Interventions: Drug: Citric acid
- Controlled group (No Intervention): No use of test meal

INTERVENTIONS:
Drug: Citric acid — Giving the citric acid (4g) solving in 200 ml of water before UBT
  Arms: Citric acid group

SUMMARY:
1. To compare the diagnostic accuracy of the 13C-Urea breath test between using the citric acid as test meal and controlled group by endoscopic biopsy methods(histology, CLOtest and H. pylori culture).
2. To compare the delta value of 13CO2 results between before and after ingestion of citric acid as test meal.

DETAILED DESCRIPTION:
1-1 Screening (visit 1, From -6 to -8 weeks) and H. pylori eradication

1. To accept the agreement, confirm inclusion/exclusion criteria, and evaluate the baseline characteristics of patients
2. H. pylori eradication

   * First eradication: PPI-based triple therapy (standard dose of PPI b.i.d., clarithromycin 500 mg b.i.d., and amoxicillin 1 g b.i.d. for 1 week), and sequential therapy (initial 5-day therapy with a combination of PPI b.i.d and amoxicillin 1g b.i.d, followed by 5 days of PPI b.i.d., clarithromycin 500mg b.i.d., and metronidazole 500mg t.i.d)
   * Rescue therapy: bismuth-containing quadruple therapy [PPI b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d.] for 1-2 weeks, or moxifloxacin-containing triple therapy (moxifloxacin 400 mg q.d., amoxicillin 1g b.i.d., and PPI b.i.d.) for 1-2 weeks.

1-2 Baseline (visit 2, 0 week): urea breath test

1. Reconfirm inclusion and exclusion criteria
2. Randomization for UBT test (citric acid group vs control group)
3. In citric acid group: taking 4 g of citric acid solving in 200 ml of water 10 minutes before UBT.
4. Perform UBT in both group

1-3) Endoscopic surveillance (visit 3, 6 or later months)

1. Endoscopic surveillance for final H. pylori status after UBT

   * Histology, CLOtest or H. pylori culture
2. Statical analysis for diagnostic accuracy of the UBT between citric acid group and controlled group: sensitivity, specificity, positive predictive value, negative predictive value, false positive rate, and false negative rate.

2. Selecting 40 patients who showed UBT result between 2.5 to 4.0 in controlled group, the investigators are planning to reperform 13C-UBT after giving citric acid as test meal.

And then, the investigators compare the change of UBT result before and after ingestion citric acid as test meal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Korean adult (Aged over 18 years)
* The Patients who diagnosed H. pylori infection and received H. pylori eradication therapy

Exclusion Criteria:

* Age under 18 years
* Patients who took any drug which could affect the study results such as proton pump inhibitor, H2 blocker, mucosal protective agents and antibiotics
* Advanced gastric cancer or other malignancy
* Abnormal liver function test or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who showed discrepant result between UBT result and endoscopic result in both citric acid group and controlled group | 6 months or later after urea breath test
  After urea breath test in the two group (citric acid group vs controlled group), endoscopic surveillance would be performed for confirmation of H. pylori status by endoscopic biopsy methods(histology, CLOtest or culture).
Compare the diagnostic accuracy which is a composite outcome measure such as sensitivity, specificity, predictive positive value and negative predictive value between citric acid group and controlled group | 6 months or later after urea breath test
  Comparing the final H. pylori status between UBT method and endoscopic biopsy methods, we will evaluate the diagnostic accuracy (sensitivity, specificity, false positive ratio, false negative ratio, positive predictive value and negative predictive value) of the UBT between using citric acid group and controlled group.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seongnam, South Korea